CLINICAL TRIAL: NCT04246463
Title: A Global Post Market Evaluation of Terumo Aortic Endovascular Grafts
Brief Title: Terumo Aortic Global Endovascular Registry
Acronym: TiGER
Status: Recruiting | Type: Observational
Sponsor: Vascutek Ltd. (Industry)
Collaborators: Bolton Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: TiGER-001
Record Dates: First submitted 2019-11-26; First posted 2020-01-29 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Abdominal Aortic Aneurysm; Thoracic Aortic Aneurysm; Surgery
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Thoracic - TEVAR
  Interventions: Device: Thoracic
- Abdominal - EVAR
  Interventions: Device: Abdominal
- Custom Device
  Interventions: Device: Custom Device
- Other indications: Isolated Iliac Artery Aneurysm (IIAA)
  Interventions: Device: Illiac Artery

INTERVENTIONS:
Device: Thoracic — Implant of a Relay stent graft system
  Groups: Thoracic - TEVAR
Device: Abdominal — Implant with an Anaconda or Treo Stent graft system
  Groups: Abdominal - EVAR
Device: Custom Device — Implant of a Fenestrated device such as Fenestrated Anaconda or Fenestrated TREO, Relay Branch or other customised device
  Groups: Custom Device
Device: Illiac Artery — Implant with an Anaconda Iliac leg only
  Groups: Other indications

SUMMARY:
Multi-arm, multi-center, open label, prospective observational registry designed to obtain safety and performance data on the use of CE marked and custom Terumo Aortic endovascular grafts.

DETAILED DESCRIPTION:
Post Market registry collecting real world, post-approval safety, performance, patient reported outcomes and health economic data on patients treated with Terumo Aortic endovascular stent-grafts in standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* • Minimum age as per local regulations

  * Indication for aortic endovascular repair with an approved or CE marked by a Regulatory body or custom-made Terumo Aortic Endovascular graft
  * Ability to provide informed consent

    o Emergent cases (typically younger patients with traumatic injuries) are not excluded if there is IRB/EC agreement to allow consent after intervention (i.e. consent to study participation, not to treatment)
  * Willingness to comply with the registry protocol
  * Willingness to adhere to follow-up visits Note: Patients currently enrolled and actively participating within the TREO registry (IP-0020-16) can have their data migrated from TREO to the TiGER registry where local EC approval has been obtained and the patient has been reconsented to TiGER for longer follow-up.

Exclusion Criteria:

* • Patient is unable or unwilling to comply with the study follow-up regime.

  * Patient is contraindicated per the IFU, or has any other medical, social or psychological problems that in the opinion of the investigator preclude them from receiving treatment as well as the procedures and evaluations pre and post procedure
  * Patient is eligible to be enrolled in or is currently actively participating in the Terumo Aortic Global FACT clinical study (FACT-001)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled under one of the following Modules Thoracic - TEVAR (Thoracic endovascular aneurysm/aortic repair) Patients requiring urgent or elective endovascular treatment of thoracic aortic aneurysm, pseudoaneurysm, dissection, penetrating aortic ulcer or intramural hematoma Abdominal - EVAR (Endovascular aneurysm/aortic repair) Patients requiring urgent or elective endovascular treatment of infrarenal abdominal aortic aneurysm.
  Custom Device - FEVAR (Fenestrated endovascular aneurysm/aortic repair) Patients with a documented thoracic or abdominal pathology suitable for elective treatment using a custom-made Terumo Aortic endovascular device.
  Other Isolated Iliac Artery Aneurysm (IIAA) Patients requiring urgent or elective endovascular treatment of isolated Iliac Artery Aneurysms (IAA)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-12-17 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Aortic Related Mortality | 30 days post implant
  Defined as any death occurring within 30 days of implant, due to rupture or following any procedure intended to treat the target lesion

SECONDARY OUTCOMES:
Technical Success | Day 0
  defined as: Successful delivery of the device through the vasculature (i.e. ability to deliver the implant to the intended location without the need for unanticipated corrective intervention related to delivery) Deployment of the endovascular stent graft in the planned location with coverage of the target lesion; Patency of the endovascular stent graft, absence of device deformations (e.g. kinks, stent eversion, mal-deployment, misaligned deployment) requiring unplanned placement of an additional device within the endovascular stent graft, and; Successful withdrawal (i.e. successful withdrawal of the delivery system, without the need for unanticipated corrective intervention related to withdrawal) Absence of Type Ia, Type Ib, Type IIIa and Type IIIb endoleak
Composite Clinical Success | 1 year
  defined as the absence of: Target lesion related mortality Target lesion aortic rupture Target lesion reintervention Occurrence of Endoleaks (Type Ia, Ib, III and IV) Loss of stent patency (>50%) Clinically significant stent graft migration (≥10mm) Stent fracture Stroke (modified Rankin Scale score of 2 or more at 90 days and an increase in at least one mRS category from an individual's pre-stroke baseline) New onset renal failure requiring dialysis Graft infection or thrombosis Where aneurysm is present Aneurysm expansion (diameter ≥5 mm, or volume ≥5%)

OTHER OUTCOMES:
Patient Outcome measure | 1 Year
  • Post-operative return to normal activities - employment, household activities, social life and hobbies (return to normal activities will be recorded at one year visit only)
Health Economics | Day 0
  The following health economic will also be summarized:
  Total procedure timea Arterial access route and type Volume of contrast media used Fluoroscopy time Image fusion technology used Magnet system used Device re-positioned Blood loss Blood transfusion required Lower limb ischemia Time in ICU/MCUb Time to hospital dischargec Complications requiring reintervention/re-hospitalisation a Time from the first break of skin to final closure (i.e., skin to skin time, percutaneous, first access to last access closure).
  b Time from the first administration of anesthesia to release from the ICU or post-anesthesia care unit providing ICU-level care. If the patient is not admitted to the ICU, this is defined as 0 hours.
  c Time from initiation of the procedure to physical discharge from the hospital.

CONTACTS AND LOCATIONS:
Locations (44):
- United States (7):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Loyola University of Chicago (Loyola), Chicago, Illinois
  - Ascension St. Vincent Heart Center, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Baylor, Scott & White Health (BSW Health), Texas City, Texas
  - University of Utah, Salt Lake City, Utah
  - Sentara Heart Hospital, Norfolk, Virginia
- Imeldaziekenhuis, Bonheiden, Belgium
- France (2):
  - Hôpital Pneumologique et Cardiovasculaire Louis-Pradel, Bron
  - CHU St Etienne, Saint-Etienne
- Germany (8):
  - Klinikum Augsburg, Augsburg
  - Evangelisches Krankenhaus Hubertus, Berlin
  - Klinikum Chemnitz, Chemnitz
  - University Heart Center Freiburg, Freiburg im Breisgau
  - Aortic Center University Hospital, Göttingen
  - Bonifatius Hospital, Lingen
  - St. Franziskus Hospital, Münster
  - University Hospital Tübingen, Tübingen
- Italy (7):
  - Policlinico Consorziale di Bari, Bari
  - Compensorio Sanitario Bolzano, Bolzano
  - Cagliari-Ospedale Brotzu, Cagliari
  - Firenze Ospedale Careggi, Careggi
  - Azienda Ospedaliera di Catania, Catania
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Maurizano Torino (turin), Turin
- Netherlands (7):
  - Vumc Amsterdam, Amsterdam
  - Rijnstate Arnham, Arnhem
  - Medisch Spectrum Twente, Enschede
  - UMC Gronigen, Groningen
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus University Medical Center, Rotterdam
  - Diakonessenhuis, Utrecht
- Portugal (3):
  - Centro Hospital Uni Lisboa Norte, Lisbon
  - Hospital de Santa Marta, Lisbon
  - CHU Sao Joao, Porto
- Spain (4):
  - Hospital Universitari Germans, Badalona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitari Valle Hebrón de Barcelona, Barcelona
  - Hospital Universitario Central de Asturias, Oviedo, Oviedo
- Switzerland (2):
  - Luzerner Kantonsspital, Lucerne
  - Civico, Ospedale Regionale, Lugano
- United Kingdom (3):
  - Hull Royal Infirmary, Hull
  - Manchester Royal Infirmary, Manchester
  - Oxford University Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Undecided